CLINICAL TRIAL: NCT02571010
Title: Pilot Study to Evaluate the Effectiveness of Somatosensory Rehabilitation of Pain by Vibrotactile Stimulation on Static Mechanical Allodynia of Less Than Three Months Duration
Brief Title: Evaluation of the Efficacy of Somatosensory Rehabilitation of Pain by Vibrotactile Stimulation on Static Mechanical Allodynia
Acronym: RESISTAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CRRF La Châtaigneraie (Other)
Collaborators: Hôpitaux Universitaires Paris Ile-de-Franc Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14RBD-RESISTAL; 2014A013 08-39 (Registry Identifier: N°IDRCB)
Record Dates: First submitted 2015-08-31; First posted 2015-10-08 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Allodynia
Keywords: static mechanical allodynia; somatosensory rehabilitation; vibrotactile stimulation
MeSH Terms: conditions — Hyperalgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vibrotactile stimulation (Experimental): Patients in this arm will have
  * treatment by medications and rehabilitation
  * treatment by vibrotactile at medical center
  * stimulation at home by soft tissue
  * non stimulation on allodynia area
  Interventions: Other: Standard Medical treatment; Device: Vibrotactile stimulation
- Sham Stimulation with Vibradol device switched off (Sham Comparator): Patients in this arm will have
  * treatment by medications and rehabilitation
  * Sham vibrotactile treatment at medical center but with Vibradol device switched off
  * abdominal breath exercises at home
  * non stimulation on allodynia area
  Interventions: Other: Standard Medical treatment; Device: Sham Stimulation with Vibradol device switched off
- Standard Medical treatment (Other): Observational group, treated as usually by medications and rehabilitation.
  Interventions: Other: Standard Medical treatment

INTERVENTIONS:
Other: Standard Medical treatment — Standard treatment with drugs and usual rehabilitation
Device: Vibrotactile stimulation — Rehabilitation by vibrotactile stimulation at medical center
  Arms: Vibrotactile stimulation
Device: Sham Stimulation with Vibradol device switched off — Sham Rehabilitation at medical center but with Vibradol device switched off
  Arms: Sham Stimulation with Vibradol device switched off

SUMMARY:
This study aims to demonstrate that somatosensory rehabilitation of pain associated with static mechanical allodynia has superior efficacy over placebo treatment as well as over spontaneous changes.

DETAILED DESCRIPTION:
This is a monocenter study. 45 patients will be enrolled in the study, allocated by randomization in 3 arms of 15 patients each.

During the 38 week duration of the study, enrolled patients will be assessed at:

* initial evaluation (first week of the study),
* intermediary evaluation for every week and every modification of intensity of pain,
* final evaluation at 10 weeks,
* follow-up evaluation at 6 months.

ELIGIBILITY:
Eligibility Criteria

1. Male or female patients aged ≥18 years;
2. Static mechanical allodynia for less than 3 months, whatever its etiology and topography;
3. Probable peripheral or central neuropathic pain or defined according to the IASP criteria;
4. Neuropathic pain diagnostic questionnaire DN4 score ≥ 4/10;
5. Chronic pain with average intensity ≥ 4/10;
6. Analgesic treatment unchanged within 15 days prior to screening, and not planned to be modified during the study;
7. Patient who can attend follow-up visits during the study;
8. Patient affiliated to a health insurance plan or entitled;
9. Patient must be able to give informed consent in accordance with ICH GCP guidelines and local legislation and/or regulations.

Exclusion Criteria:

1. Patient with neuralgia (spontaneous pain) with or without allodynia;
2. Patient not able to participate actively to the rehabilitation exercises for physical reason, cognitive reason (ability to understand instructions) or behavioural reason (e.g. addiction...);
3. Patient with complex regional pain syndrome (type I);
4. Patients for whom cares cannot avoid any touch with allodynia area;
5. Patient previously treated by a transcutaneous electrical nerve stimulation (TENS);
6. Prior treatment by somatosensory rehabilitation;
7. Duration of stay in the medical center < 11 weeks;
8. Patient with cognitive disorder;
9. Allodynia area of the patient presenting with conditions not recommended for vibrotactile stimulation: wound, unhealed nerve suture, recent skin transplantation, fragile organ such as eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Change of baseline in reduction of surface of allodynia area | At baseline, each week during the 10 week treatment period and at 6 months
  Evaluate by the 15 g mono filament (Allodynographie) the reduction of surface of allodynia area

SECONDARY OUTCOMES:
Change of baseline in reduction of pain | At baseline, at each week, at 10 weeks and at 6 months
  Reduction of pain will be evaluated by QDSA questionnaire.
Change of baseline in reduction of allodynia intensity | At baseline, at each week, at 10 weeks and at 6 months
  Reduction of allodynia intensity will be measured with the method with the colors
Change of baseline of patient's satisfaction with regard to received care | At baseline, at each week, at 10 weeks and at 6 months
  Patient's satisfaction with regard to pain relief will be evaluated by VAS
Analgesics consumption | At 6 months
  Amount of analgesic drugs
Afterglow effect | At 6 months
  An evaluation of static mechanical allodynia in surface and intensity at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rania Belmahfoud, MD, Study Chair — CRRF La Chataigneraie Convention; Valérie Zingale, Study Director — CRRF La Chataigneraie Convention
Locations (1):
- CRRF La Chataigneraie Convention, Paris, Île-de-France Region, France